CLINICAL TRIAL: NCT05998460
Title: Glucose-Guided Eating to Reduce Chronic Disease Risk: a Pilot Study
Brief Title: Glucose-Guided Eating Pilot
Acronym: GET CHARGED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00006573
Record Dates: First submitted 2023-07-21; First posted 2023-08-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-06

CONDITIONS: Postmenopausal; Prediabetes; Adolescent and Young Adult (AYA) Cancer Survivors
MeSH Terms: conditions — Prediabetic State | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GGE with CGM (Experimental): Participants randomized to the Glucose-Guided Intervention will be trained to align their mealtimes with a personalized glucose threshold monitored using continuous glucose monitoring (CGM) and the GGE study app.
  Interventions: Behavioral: Glucose-Guided Eating with CGM; Other: CGM only
- CGM only (Active Comparator): Participants randomized to the control arm will only wear a CGM.
  Interventions: Other: CGM only

INTERVENTIONS:
Behavioral: Glucose-Guided Eating with CGM — The GGE intervention consist of up to four weeks of training to learn to eat when glucose levels are at or below their usual fasting level. Specifically, participants following GGE will self-monitor their glucose levels with an unblinded CGM while using a mobile app (GGE app) that will provide feedback on whether or not to eat. At desired mealtimes participants will enter their current glucose level, rate their perceived hunger, and label the type of hunger they are experiencing (physical, emotional, sensory and practical). Participants following GGE will be instructed by the app to eat when two conditions are met: (a) the desire to eat arises and (b) their glucose levels are at or below a personalized threshold. During the training period, participants are meant to associate feelings of perceived hunger with fasting glucose levels (i.e., physical hunger). After the training period, participants continue to follow GGE without CGM or use of the app.
  Arms: GGE with CGM
Other: CGM only — Comparator participants will use unblinded CGM for up to 4 weeks without the use of the GGE app or any other dietary recommendations.

SUMMARY:
This is a single center, parallel-arm randomized controlled pilot study that aims to examine the feasibility and acceptability of the glucose-guided eating (GGE) mobile app and intervention in two populations at risk of chronic disease (postmenopausal women with prediabetes and AYA cancer survivors).

DETAILED DESCRIPTION:
The primary objectives of the study are to (1) test the feasibility and acceptability of the GGE intervention and companion GGE mobile app and (2) quantify the preliminary effect of GGE on 12-week changes in insulin resistance (IR) and body weight.

The secondary objectives of the study are to (1) collect preliminary data on hypothesized mechanisms linking GGE to IR and (2) explore the durability of intervention effects on 24-week changes in body weight.

ELIGIBILITY:
Inclusion Criteria:

All:

1. Self-reported height and weight that is consistent with a BMI ≥ 27 kg/m2
2. Willing to use a continuous glucose monitor
3. Own smartphone that is compatible with Dexcom CGM.
4. Willingness to commute to GUMC for in-person study visits
5. No active cancer (except for nonmelanoma skin cancer)
6. Less than 5 lbs. weight change in previous 3 months
7. Proficient in speaking and reading English

   Postmenopausal women with pre-diabetes:
8. Age 18 years and older
9. Diagnosed as having prediabetes.
10. HbA1c (within 3 months) between 5.7% and 6.4%
11. Postmenopausal (defined as reporting no menstrual period for ≥1 year or a reported history of a total abdominal hysterectomy with oophorectomy)

    AYA cancer survivors:
12. Current age 21-39 years
13. Previously diagnosed with cancer, with all cancer-related diagnosis chemotherapy and/or radiation completed at least 6 months previously

Exclusion Criteria:

1. Unable or unwilling to provide informed consent
2. Clinical history of type 1 or type 2 diabetes
3. Currently receiving anti-diabetics (e.g., insulin, GLP1), oral hypoglycemic agent (e.g., metformin), oral corticosteroids, oral glucocorticoids, beta blockers, hydroxyurea, atypical antipsychotic agents (i.e., Olanzapine, Aripiprazole) or systemic progestin-only contraceptives
4. Current or past history of an eating disorder
5. Self-identify as an overnight eater (defined as eating main meals between 9pm-5am)
6. Have any contraindications for CGM, including: severe allergy to surgical adhesive, being on dialysis, receiving diathermy treatment, or scheduled CT scan or MRI during wear period
7. Growth hormone deficiency, hypoadrenal function, or hypopituitary function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-02 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Population-specific accrual | Week 0
  Population-specific accrual will reflect rates of study enrollment and will be defined as number of participants consented to the number of individuals who are determined to be eligible.
Population-specific retention rates | Week 12
  Population-specific retention rates will reflect the proportion of enrolled participants who complete the study.
GGE app usability | Week 12
  The app usability will be assessed using the 10-item System Usability Scale. SUS scores have a range of 0 to 100 with 100 representing greatest usability.
GGE intervention acceptability | Week 12
  GGE intervention acceptability will be assessed with a study specific survey (collected from participants randomized to the GGE intervention only).
GGE adherence | Weeks 1-4
  GGE adherence will be quantified as percent of reported eating events occurring at or below personalized glucose thresholds/personalized average fasting glucose levels that is collected using the GGE app (collected from participants randomized to the GGE intervention only-during use of the GGE app only).

SECONDARY OUTCOMES:
Changes in body weight | Weeks 0-12 and Weeks 12-24
  Changes in body weight will be measured using calibrated digital scales (measured in kilograms).
Changes in insulin resistance (HOMA-IR) | Weeks 1-12
  Changes in insulin resistance will be measured as homeostatic model assessment for insulin resistance (HOMA-IR). It will be computed from fasting insulin and fasting glucose (fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5).
Changes in glycemic variability | Weeks 1-12
  Changes in glycemic variability will be assessed from CGM data using the freely accessible EasyGV software available from the University of Oxford (https://www.phc.ox.ac.uk/research/resources/easygv).
Changes in oxidative stress | Weeks 1-12
  Changes in oxidative stress will be measured as 8-isoprostane from spot urine.
Changes in the soluble receptor for advanced glycation end-products (sRAGE) | Weeks 1-12
  Changes the sRAGE was measured in serum by ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Schembre, Principal Investigator — Georgetown's Lombardi Comprehensive Cancer Center; Nina Kadan-Lottick, Principal Investigator — Georgetown's Lombardi Comprehensive Cancer Center

IPD SHARING:
Plan to Share IPD: Yes
The investigators intend to publish the protocol in a manuscript and share the IPD through an appropriate free access data repository.
Time Frame: Within 1 year of study completion.
Access Criteria: Shared IPD will be available via freely accessible data registry.

REFERENCES:
- [Background] Schembre SM, Jospe MR, Giles ED, Sears DD, Liao Y, Basen-Engquist KM, Thomson CA. A Low-Glucose Eating Pattern Improves Biomarkers of Postmenopausal Breast Cancer Risk: An Exploratory Secondary Analysis of a Randomized Feasibility Trial. Nutrients. 2021 Dec 16;13(12):4508. doi: 10.3390/nu13124508. PMID 34960058
- [Background] Schembre SM, Jospe MR, Bedrick EJ, Li L, Brewster AM, Levy E, Dirba DD, Campbell M, Taylor RW, Basen-Engquist KM. Hunger Training as a Self-regulation Strategy in a Comprehensive Weight Loss Program for Breast Cancer Prevention: A Randomized Feasibility Study. Cancer Prev Res (Phila). 2022 Mar 1;15(3):193-201. doi: 10.1158/1940-6207.CAPR-21-0298. PMID 34893531